CLINICAL TRIAL: NCT04208919
Title: Safety and Preliminary Efficacy of Delayed Donor-derived Regulatory Dendritic Cell (DCreg) Infusion and Immunosuppression Withdrawal in Living Donor Liver Transplant (LDLT) Recipients
Brief Title: Delayed Infusion of DCreg in Living Donor Liver Transplantation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Angus W. Thomson PhD DSc (Other)
Responsible Party: Sponsor-Investigator, Angus W. Thomson PhD DSc, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY20010215
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Living Donor Liver Transplantation
Keywords: Regulatory Dendritic Cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DCreg Prior to Weaning (Experimental): Regulatory dendritic cells that were derived from the recipient's liver donor will be infused into the recipient one week prior to the initiation of immunosuppression weaning.
  Interventions: Biological: Donor-derived DCreg

INTERVENTIONS:
Biological: Donor-derived DCreg — Regulatory dendritic cells that were prepared from a donor leukapheresis will be infused into liver transplant recipients 7 days prior to the start of immunosuppression weaning.

SUMMARY:
Phase I/II, single center, prospective, open-label, non-controlled, non-randomized, interventional, cohort study in which low risk living donor liver transplant (LDLT) recipients who are between 1 and 3 years after transplantation and meet specific criteria (no positive crossmatch, no clinically treated rejection within 2 years preceding enrollment, permissive liver function tests (LFTs) within 30 days preceding enrollment, no prior liver biopsy showing significant fibrosis or ductopenia*) will be enrolled and will undergo a protocol liver biopsy unless they have had a permissive liver biopsy** within 90 days of anticipated immunosuppression weaning. Those patients with permissive liver biopsy** will then receive a single infusion of donor-derived DCreg and will remain on their current standard of care (SOC) immunosuppression. One week after DCreg infusion, immunosuppression weaning will be initiated. Recipients will be slowly weaned off immunosuppression. Successfully weaned participants who remain rejection-free will undergo 3 years of follow-up after the last dose of immunosuppression. They will undergo a liver biopsy at 1 yr and 3 yrs after immunosuppression withdrawal. Participants who are removed from the study protocol at any time will return to standard of care but will continue to be followed by the study team and will undergo a liver biopsy at the end of the study.

* Permissive LFTs are defined as ALT, AST and total bilirubin < 2.5 times the upper limit of normal.

**A permissive biopsy is based on 2016 Comprehensive Update of the Banff Working Group on Liver Allograft Pathology (the criteria detailed in Table 8, Demetris et al. 2016).

DETAILED DESCRIPTION:
Long-term immunosuppression after solid organ transplantation is associated with life-threatening side effects that include infection, malignancy, diabetes and increased risk of cardiovascular disease. In addition, use of calcineurin inhibitors (CNI) causes nephrotoxicity and a significant rate of chronic renal insufficiency (CRI) at 5 years after orthotopic liver transplantation (OLT). Many patients with CRI after OLT require renal replacement therapy (dialysis or renal transplantation) and are at increased mortality risk. A large study based on the Scientific Registry of Transplant Recipients (SRTR) and the Centers for Medicare and Medicaid Services (CMMS) ESRD Program database showed an ESRD incidence of 15 per 1000 patient years, implying that in 20 years, ~30% of patients require renal replacement therapy. Patients demonstrating progressive loss in functional nephron mass are also at risk of progressing to chronic kidney disease (CKD), which is known to confer > 4 fold increase in mortality risk. Immunosuppression (CNI) withdrawal, particularly before significant renal injury has set in, may preserve renal function and prevent morbidity and mortality associated with CKD/CRI and renal replacement therapy. Immunosuppression withdrawal may also mitigate the increased risk of infection, malignancy, diabetes, and cardiovascular disease directly associated with conventional immunosuppressive medications.

Our goal is to develop a novel, safe cell therapy approach that, when used in liver transplantation would facilitate the safe complete withdrawal of immunosuppression without jeopardizing allograft function or histology. Recent evidence suggests that, by exploiting inherent mechanisms of immune regulation, it may be possible to achieve this goal. Rare, naturally-occurring regulatory immune cells, either innate or adaptive, critically regulate immunity, promote antigen (Ag)-specific T cell hyporesponsiveness and prevent adverse immune reactions in the healthy steady-state. In addition to Treg, being evaluated for cell-based therapy in organ transplantation, a compelling rationale has emerged for clinical testing of regulatory DC modified ex vivo to promote their regulatory properties (DCreg). Thus, in rodents, infusion of donor-derived DCreg before transplantation, including their combination with conventional IS, promotes indefinite (> 100 day) organ allograft survival. There is also evidence that infusion of donor- or recipient- derived DCreg post-transplant can promote indefinite allograft survival. More importantly and uniquely, using a robust, clinically-relevant, non-human primate (NHP) model with minimal IS, we have shown that infusion of DCreg, one week before transplantation, significantly and safely prolongs renal allograft survival, with no evidence of host sensitization. Equally significant, is our demonstration that prolongation of allograft survival is associated with selective attenuation of donor-reactive Tmem responses, an important barrier to improving long-term graft survival and achieving operational tolerance.

Development of safe and effective approaches that improve long-term graft survival while reducing the burden of conventional immunosuppressive drugs, will have a significant impact on the health, as well as costs, of thousands of organ transplant recipients. Extensive pre-clinical studies conducted by Dr. Thomson (IND Sponsor) and others in rodents and humanized mouse models are persuasive regarding the potential of regulatory immune cell therapy to enhance long-term allograft survival and in many instances, promote donor-specific tolerance. The case for evaluation of DCreg generated ex vivo is particularly compelling. First, DC are inherently tolerogenic, uniquely well-equipped, professional Ag-presenting cells (APC) that potently regulate innate and adaptive immunity. Second, in many animal studies, DCreg adoptively transferred to allograft recipients before or after transplant induce Ag-specific tolerance and promote indefinite graft survival. Moreover, this therapeutic effect does not appear to depend on the in vivo persistence of intact DCreg. Independence of efficacy and underlying regulatory mechanisms on persistence of intact donor DCreg may be a distinct advantage over other cell therapy approaches, where costly repeated infusion of large numbers of cells and their sustained viability/stability/replication may be required to achieve a therapeutic effect. Third, an important attribute of DCreg is their ability to regulate preformed Tmem responses, that, due to molecular mimicry, cross-react with HLA Ags [66], representing a major barrier to long-term graft survival in humans. Fourth, in normal humans, adoptive transfer of monocyte-derived DCreg induces Ag-specific inhibition of effector T cell function. Fifth, using minimal IS in a robust, NHP model, we have reported that a single infusion of 3.5-10.106/kg donor-derived DCreg pre-transplant safely prolongs renal allograft survival, without host sensitization. Importantly, this effect is associated with attenuation of donor-specific, alloreactive Tmem responses.

The DCreg approach could be readily applied in the clinic since a single infusion of a relatively small number of DCreg (3.5-10.106/kg) in NHP is sufficient to achieve a salutary therapeutic effect. Therefore, neither expensive expansion of the cell product over several weeks (compared with Treg), nor repeated infusion appears necessary. It is also likely that DCreg will have broader clinical application to encompass recipients of organ transplants from deceased donors as rodent studies have shown that delay of DCreg infusion to 7 or 14 d after transplant is still effective in prolonging graft survival and promoting tolerance, providing ample time to prepare DCreg from deceased donors.

The possibility that DCreg administration could enable early withdrawal of immunosuppression (< 3 years) after liver transplantation carries the potentially great advantage of sparing patients the cardiovascular, infectious, neoplastic, and renal side effects of long-term immunosuppression, particularly with CNI. Liver transplantation provides a particular opportunity to achieve this goal because liver grafts are more tolerated by the recipient's immune system than other solid organ grafts, with immunosuppression withdrawal possible in ~20% of patients overall (in the absence of any experimental, immunomodulatory therapy) compared to <5% in renal transplant recipients. Increasing the proportion of liver transplant recipients who can be withdrawn from immunosuppression through the administration of DCreg around the time of transplantation could reap significant health benefits to this patient population.

ELIGIBILITY:
Inclusion Criteria:

Donor

1. Able to understand and provide informed consent
2. Male or female age 18 or older at the time of enrollment
3. Have no contraindication to leukapheresis
4. For females of childbearing potential, a negative urine or serum pregnancy test
5. No live vaccines within 12 weeks prior to leukapheresis
6. Negative health history for risk factors related to Creutzfeldt-Jakob disease
7. Negative for West Nile Virus(a)
8. Negative for HIV (5th generation Test and NAT), HTLV-1, HTLV-2;(a)
9. Negative for hepatitis C (antibody and NAT), hepatitis B (surface antigen and NAT)(a)

   1. does not preclude donors from undergoing leukapheresis but cells may not be infused into recipient.

Recipients

1. Low risk LDLT recipients, irrespective of gender, race, or ethnic background. Low risk is defined by absence of exclusion criteria (below).
2. Age 18 or older at the time of enrollment
3. Underwent de novo (first) liver transplant 1 to 3 years prior to enrollment
4. Female subjects of childbearing potential must have a negative pregnancy test upon study entry.
5. Agreement to use contraception; according to the FDA Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective. Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from this list to be used from the time that study treatment begins until 1 year after completion of immunosuppression withdrawal.

Exclusion Criteria:

Recipients

1. History of positive crossmatch (performed prior to transplant)
2. Clinically treated rejection episode within 2 years prior to enrollment
3. Non-permissive LFTs within past 1 month
4. Repeat liver transplant
5. Prior other solid organ transplant
6. Significant co-morbid conditions such as severe heart or lung disease
7. Following etiology of liver disease: Primary Sclerosing Cholangitis (PSC), autoimmune, Primary Biliary Cirrhosis (PBC)
8. If prior history of Hepatitis B or C (HBV or HCV) infection, Hepatitis B or C Virus (HBV or HCV) viral load positive at the time of enrollment (successfully treated HBV or HCV patients are not excluded)
9. Positive antigen-antibody immunoassay for HIV-1/2
10. Any prior biopsy showing significant fibrosis or ductopenia.
11. Any medical condition that the investigator deems incompatible with participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of recipients who experience CTCAE Grade 4 or higher infusion reaction | 1 day
  Safety will be determined by assessing the proportion of subjects who experience CTCAE Grade 4 or higher infusion reaction
The proportion of recipients who experience CTCAE Grade 4 or higher infection | 4 years
  Safety will be determined by assessing the proportion of subjects who experience CTCAE Grade 4 or higher infection
The proportion of recipients who experience experience malignancy other than non-melanoma skin cancer or HCC recurrence | 4 years
  Safety will be determined by assessing the proportion of subjects who experience malignancy other than non-melanoma skin cancer or HCC recurrence
The proportion of recipients who experience rejection resulting in recipient death or retransplantation | 4 years
  Safety will be determined by assessing the proportion of subjects who experience rejection resulting in recipient death or retransplantation
The proportion of recipients who experience biopsy-proven severe acute rejection | 4 years
  Safety will be determined by assessing the proportion of subjects who experience biopsy-proven severe acute rejection
The proportion of recipients who experience any grade chronic rejection | 4 years
  Safety will be determined by assessing the proportion of subjects who experience any grade chronic rejection
The proportion of recipients who experience non-surgical graft loss | 4 years
  Safety will be determined by assessing the proportion of subjects who experience non-surgical graft loss
The proportion of recipients who die | 4 years
  Safety will be determined by assessing the proportion of subjects who die
Preliminary Efficacy of using DCreg therapy to facilitate immunosuppression weaning | 2 years
  Proportion of patients able to achieve immunosuppression withdrawal with operational tolerance 1 year after complete immunosuppression cessation based on specific liver biopsy criteria

SECONDARY OUTCOMES:
Donor Specific Antigen (DSA) levels | 4 years
  DSA levels early (<4 wks) and late (>4 wks) after DCreg infusion
Change in renal function | Change from baseline to 36 months post-weaning
  Change in renal function (defined as estimated GFR calculated by CKD-EPI: http://www.qxmd.com/calculate-online/nephrology/ckd-epiegfr) between time of enrollment and 1 year following immunosuppression weaning will be calculated.
Change in Quality of Life as measured by the Short Form 36 (SF-36) | Change from baseline to 36 months post-weaning
  This 36-item questionnaire measures general health-related quality of life, with scores ranging from 0 to 100; a higher score indicates a better health state. Two component scores, Mental Component Score and Physical Component Score, are derived from 8 domain scores. The 8 domains [US Population Means] are: 1) Physical Functioning [84.2], 2) Role-physical [81.0], 3) Bodily Pain [75.2], 4) General Health [72.0], 5) Vitality [60.9], 6) Social Functioning [83.3], 7) Role-emotional [81.3], and 8) Mental Health [74.7]
Change in cardiovascular risk factors | Change from baseline to 36 months post-weaning
  Cardiovascular factors assessed include incidence of hypertension necessitating medication, post-transplantation diabetes, hyperlipidemia, hypercholesterolemia as documented from medical record review at yearly post-transplant visits.

CONTACTS AND LOCATIONS:
Overall Officials: Abhinav Humar, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No